CLINICAL TRIAL: NCT01224496
Title: Traditional Chinese Medicine in the Supportive Management of Anaemic and Cytopenic (Leukopenia, Thrombocytopenia) Haematological Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Shanghai Yueyang Integrated Medicine Hospital (Other); Singapore Bao Zhong Tang TCM Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SHF/TCM002/2008
Record Dates: First submitted 2010-10-03; First posted 2010-10-20 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Myelodysplastic Syndrome (MDS); Aplastic Anaemia (AA); Myelofibrosis (MF); Thalassemia Intermedia
Keywords: Chronic cytopenic haematological diseases; Chinese herbal concoction; Supportive management
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Aplastic; Primary Myelofibrosis; beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with Chinese herbal concoction (Experimental): Patients must have a marrow study to confirm diagnosis of MDS, AA or MF. MDS is classified according to the WHO criteria and scored according to IPSS. The AA group is further classified into AA, SAA or VSAA . MF is defined by the Italian criteria and risk stratified by the Lilles Scoring system. Diagnosis of thal intermedia and major is based on previously done Hb electrophoresis and severity of disease is assessed by degree of anaemia.and frequency of blood transfusions
  TCM diagnosis: Syndrome differentiation according to TCM theory will be assessed as a baseline by experienced TCM collaborators and classified into one of the few defined syndromes as follows
  1. Yin deficiency of spleen and kidney
  2. Yang deficiency of spleen and kidney
  3. Deficiency of both Yin and Yang
  4. Stagnation of dampness and poison in the blood
  5. Excessive heat and poison
  Interventions: Drug: Chinese herbal concoction twice a day for 6 months

INTERVENTIONS:
Drug: Chinese herbal concoction twice a day for 6 months — Definition of each TCM syndrome is based on TCM theory. Formulation composition is based on each defined TCM syndrome with addition or removal of herbs as indicated by the patient's manifestation

SUMMARY:
The purpose of this study is to study the efficacy of Traditional Chinese Medicine (TCM) on anaemic and cytopenic haematological disorders including myelodysplastic syndrome (MDS), aplastic anaemia (AA), myelofibrosis (MF) and thalassemia intermedia who do not have or did not respond to available treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of MDS, AA, MF or thal based on currently recognized diagnostic criteria.
2. Explored or undergone established therapies eg haemopoietic stem cell transplant, immunosuppressive therapy, chemotherapy, growth factors, thalidomide, hypomethylating agent or androgens, and (a) are deemed not suitable, or (b) refuse or (c) have failed therapy
3. A preceding follow up period (without or with treatment) of 2-4 months as baseline (depending on the severity of cytopenia) before being enrolled into this study
4. Understand the trial nature of this treatment, agree to be compliant to medication, do not self medicate and have signed informed consent
5. Agreeable to regular blood tests and follow up marrow study as listed in schedule

Exclusion Criteria:

1. Life expectancy of shorter than one year
2. Significant organ failure including the following
3. Renal impairment with Cr above 200umol/L
4. Liver impairment with serum bilirubin > 2x upper limits or transaminase >3x upper limits
5. Escalation of treatment of introduction of new agents including growth factors, thalidomide, hypomethylating agents, immunosuppressive therapy or androgens once started on treatment with TCM is not allowed. Continuation of current therapy at same or lower doses is allowed
6. Women during pregnancy or lactation.

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 6 months
  The following parameters will be monitored serially
  1. symptoms : ie reflection of any subjective symptoms that may be due to the treatment
  2. Serial biochemistry ( urea, electrolyte, creatinine, liver function test ) will be done at baseline, one week into the study and then every 7-8 weekly till end of the 6 months. This will monitor for any organ toxicity

SECONDARY OUTCOMES:
Quality of life | 6 months
  Quality of life (QOL) will be measured based on the EORTC QLQ C30. THis will be taken at enrolment and at 2 monthly intervals
Haematological improvement | 6 months
  The haematological response crietria is based on those published as follows
  For MDS : Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood 2000 Dec 1;96(12):3671-4.
  For MF : Response criteria for myelofibrosis with myeloid metaplasia: results of an initiative of the European Myelofibrosis Network (EUMNET). Blood 2005 Oct 15;106(8):2849-53.
  For AA : Aplastic Anemia, Pathophysiology and Treatment. Cambridge: Cambridge University Press; 2000.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Linn YC, Lu J, Lim LC, Sun H, Sun J, Zhou Y. Traditional Chinese herbal medicine in the supportive management of patients with chronic cytopaenic marrow diseases -- a phase I/II clinical study. Complement Ther Clin Pract. 2011 Aug;17(3):152-6. doi: 10.1016/j.ctcp.2011.01.004. Epub 2011 Feb 17. PMID 21742281